CLINICAL TRIAL: NCT01785264
Title: Non-operative Treatment of Acute Achilles Tendon Ruptures Versus Open and Mini-invasive Surgery: A Prospective Randomized Trial.
Brief Title: Treatment Results After Acute Rupture of the Achilles Tendon.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Oslo University Hospital (Other); Sykehuset Ostfold (Other); Vestre Viken Hospital Trust (Other); Hjelp24 (Other)
Responsible Party: Principal Investigator, Stale Bergman Myhrvold, Consultant orthopedic surgeon, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012/530/REK; 2013005 (Other: The Norwegian Regional Health Authorities)
Record Dates: First submitted 2013-01-28; First posted 2013-02-07 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Rupture of Achilles Tendon
Keywords: Achilles; Tendon; Rupture; Acute; Treatment; Outcome measure
MeSH Terms: conditions — Rupture | interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open surgery (Active Comparator): Treatment is divided into three arms, and patients between 18 and 60 years of age sustaining first time achilles tendon ruptures will be invited to participate. All three groups will have identical rehabilitation protocol. Open surgical repair is done through a 10 cm longitudinal incision, through the fascia curries and the paratenon. After necessary revision of the injure site, the tendons ends is sutured with a double layer, three knot, Krakow whip suture technique. 5 to 10 degrees of overcorrection compared to the uninjured side is endeavored. The paratenon is sewn as much as possible back over the injure site and suture material. The fascia is sutured and then continuous lying mattress skin suture.
  Interventions: Procedure: Non-operative treatment; Procedure: Open surgery; Procedure: Mini-invasive surgery
- Non-operative treatment (Active Comparator): Non-operative treatment starts with casting the ankle in equinus position. The rest of the treatment from there on will be identical to the two other arms: Minimal invasive and open surgery. Casting lasts for 2 weeks for all three arms.
  Interventions: Procedure: Non-operative treatment; Procedure: Open surgery; Procedure: Mini-invasive surgery
- Mini-invasive surgery (Active Comparator): Patients allocated to mini-invasive treatment will (as patients treated with open surgery) be operated within 7 days from injury with the technique developed by Dr Amlang and Prof Zwipp in Dresden. Patients in all three arms will have an active, early weight bearing rehabilitation protocol.
  Interventions: Procedure: Non-operative treatment; Procedure: Open surgery; Procedure: Mini-invasive surgery

INTERVENTIONS:
Procedure: Non-operative treatment — All patients included in the study will be immobilized in equinus position for the first two weeks using a below-the-knee cast. Following the first two weeks the cast is replaced with a brace that will be used for additional six weeks during which the ankle angle will be adjusted from 3 heel-lifts to none. Patients randomized to non-operative treatment will have a cast applied within 3 days from injury.
Procedure: Open surgery — All patients included in the study will be immobilized in equinus position for the first two weeks using a below-the-knee cast. Following the first two weeks the cast is replaced with a brace that will be used for additional six weeks during which the ankle angle will be adjusted from 3 heel-lifts to none.
Procedure: Mini-invasive surgery — We will use the technique developed by Dr. Amlang and Professor Zwipp from Dresden, Germany. They have developed a protocol of mini-invasive surgery using specially adapted proprietary instruments.
  All patients included in the study will be immobilized in equinus position for the first two weeks using a below-the-knee cast. Following the first two weeks the cast is replaced with a brace that will be used for additional six weeks during which the ankle angle will be adjusted from 3 heel-lifts to none.

SUMMARY:
To compare the end-results of three different methods of treatment of acute achilles tendon ruptures, it is necessary to establish identical rehabilitation protocols. Traditionally, early mobilization has been reserved for patients treated surgically and this may have unintentionally skewed treatment results. The investigators have therefore designed a prospective randomized trial performed as collaboration between Akershus University Hospital (Ahus), Oslo University Hospital (The Emergency Department), Østfold Hospital (Fredrikstad) and Drammen Hospital. The four institutions were chosen because of their geographical proximity and because they jointly have a substantial catchment area. Treatment is divided into three arms, and patients between 18 and 60 years of age sustaining first time achilles tendon ruptures will be invited to participate.

DETAILED DESCRIPTION:
Patients are randomized to either surgery or non-operative treatment. Surgery will be performed by open technique or by using a mini-invasive approach. Open surgery remains widespread and arguably the best documented treatment, however mini-invasive surgery is also included because of its potential to lessen the risk of wound complications. Michael Amlang and Hans Zwipp at the University of Dresden represent some of the leading foot- and ankle surgeons in Europe. They and their co-workers have developed a protocol for mini-invasive surgery using specially adapted proprietary instruments. Michael Amlang visited Ahus in 2012 teaching the general principles of the Dresden mini-invasive treatment. To ensure optimal and reproducible results, surgeons participating in the study must master both techniques.

All patients included in the study will be immobilized in equinus position for the first two weeks using a below-the-knee cast. Following the first two weeks the cast is replaced with a brace maintaining ∼12° plantar flexion (three heel lifts). We have chosen to use standardized heel lifts because it eases weightbearing compared to a hinged brace. After two weeks (four weeks from injury) the ankle position is adjusted to ∼8° plantar flexion (two heel lifts) and following additional two weeks the ankle position is adjusted to ∼4° plantar flexion (one heel lift). The last week of the orthosis treatment the heel lift is completely removed. Hence, the brace is retained for a total of six weeks, and patients are allowed full weight bearing as tolerated during the entire time period. The brace is worn day and night for the first two weeks, but is removed during nighttime for the last four weeks. Importantly, the immobilization regimen is identical for all three-treatment groups. To ensure identical rehabilitation following immobilization, physical therapy has to adhere to a standardized protocol supervised by an experienced physiotherapist at the Norwegian Sport Medicine Clinic (NIMI).

The defined endpoint is treatment results evaluated by the Achilles tendon Total Rupture Score (ATRS). This is a patient-centered self-reporting instrument with good reliability, validity and sensitivity. Furthermore, ATRS will be combined with SF36, another commonly used self-reporting instrument. Pain is evaluated by a visual analogue scale (VAS). Functional results are evaluated by The MuscleLab measurement system (Ergotest Innovation, Porsgrunn, Norway). The system consists of two different jump tests (drop counter-movement jump and hopping), two different strength tests (concentric heel rise and eccentric-concentric heel rise) and one muscular endurance test (standing heel rise) and the system has been shown to be both valid and reliable assessing lower leg function in patients with Achilles tendinopathy. We will also measure dorsiflexion and plantarflexion range of movement (ROM) as well as the circumference of the calf, all widely used endpoints in similar studies. Secondly, we want to compare the risk of complications such as infections and reruptures. The patients are examined at baseline and after 6 and 12 months. Since there are only minor functional improvements after 12 months, we do not plan any later follow-up as part of the main project. The 6 and 12 months examinations will be completed at the Norwegian Sport Medicine Clinic (NIMI), these examinations are blinded and performed by two physiotherapists who have not been taking part in the study prior to final follow-up. Patients will be wearing knee socks to hide potential scar tissue.

Although the minimum clinically important difference in ATRS score has yet to be determined, Carmont and coworkers have shown that 7 points represent the smallest detectable change. Moreover, a study by Metz et al. found that patients with reruptures of the achilles tendon presented on average 18 points lower scores whereas patients with injuries of the sural nerve or superficial wound infections presented scores 10 and 9 points lower than average, respectively. In order to detect a difference of 7 points in ATRS score with 80% power there must be 160 patients in each group. Power calculations are based on one-way ANOVA analyses assuming a common standard deviation of 20. This concomitantly allows us to detect differences as low as 8 % with respect to complications. This is of pivotal importance since assessing the risk of reruptures is essential when establishing treatment recommendations. We therefore plan to include a total of 530 patients allowing for expected loss during follow-up. Ahus, The Emergency Department of Oslo University Hospital, Drammen and Fredrikstad Hospitals have a catchment area of nearly 1.3 million people and treats in excess of 300 achilles tendon ruptures annually. This allows for completion of the inclusion period within three years. In our view, this is the first study to include a sufficient number of patients to detect lesser, but yet important differences, and the results will be published in a suitable international peer-reviewed journal.

The prospective randomized trial embodies many different disciplines and will spur off follow-up studies. As part of the main project we will conduct a treatment-cost analysis in relation to individual results. We will also perform an investigation based on ultrasound grading of Achilles tendon ruptures according to a classification system established by Michael Amlang and colleagues. Previous studies have provided evidence suggesting that treatment results may depend on the extension of the injury, and that treatment recommendations should be based on type of rupture sustained. This is of particular interest as it may facilitate individualized treatment. Together with the prospective randomized trial and the treatment-cost analysis, the ultrasound investigation will constitute the core of the Doctor of Philosophy (PhD) project.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 60 years of age sustaining first time achilles tendon ruptures will be invited to participate.
* The injury must be addressed with a below the knee cast in equinus position within 3 days from injury.
* The operations must be carried out within 7 days from injury.

Exclusion Criteria:

* Age below 18 or above 60 years
* The use of quinolone antibiotics within 6 months prior to injury
* Former achilles tendon injury on either side
* Steroid injections close to the achilles tendon the last 6 months
* The use of systemic steroids (prednisolon)
* Diabetes mellitus
* Dependent on walking aids
* Not able to undergo the rehabilitation protocol
* Not willing to perform the controls on the hospitals and examinations at NIMI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 530 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The defined endpoint is treatment results evaluated by the Achilles tendon Total Rupture Score (ATRS) at 12 month follow-up examination. | The patients are examined at baseline and after 6 and 12 months.
  The defined endpoint is treatment results evaluated by the Achilles tendon Total Rupture Score (ATRS). This is a patient-centered self-reporting instrument with good reliability, validity and sensitivity. Furthermore, ATRS will be combined with SF36, another commonly used self-reporting instrument. Pain is evaluated by a visual analogue scale (VAS). Functional results are evaluated by The MuscleLab measurement system (Ergotest Innovation, Porsgrunn, Norway). We will also measure dorsiflexion and plantarflexion range of movement (ROM) as well as the circumference of the calf, all widely used endpoints in similar studies.

SECONDARY OUTCOMES:
Risk of complications such as infections and reruptures within 12 months after initiation of treatment. | The patients are examined at baseline and after 6 and 12 months.
  Secondly, we want to compare the risk of complications such as infections and reruptures. The patients are examined at baseline and after 6 and 12 months. Since there are only minor functional improvements after 12 months, we do not plan any later follow-up as part of the main project. The 6 and 12 months examinations will be completed at the Norwegian Sport Medicine Clinic (NIMI), these examinations are blinded and performed by two physiotherapists who have not been taking part in the study prior to final follow-up. Patients will be wearing knee socks to hide potential scar tissue.

OTHER OUTCOMES:
SF36 after 12 months after initiation of treatment. | Baseline, 6 and 12 months
  ATRS will be combined with SF36, another commonly used self-reporting instrument. Pain is evaluated by a visual analogue scale (VAS). Functional results are evaluated by The MuscleLab measurement system (Ergotest Innovation, Porsgrunn, Norway). We will also measure dorsiflexion and plantarflexion range of movement (ROM) as well as the circumference of the calf, all widely used endpoints in similar studies.

CONTACTS AND LOCATIONS:
Overall Officials: Ståle B Myhrvold, MD, Principal Investigator — University Hospital, Akershus; Sigurd E Hoelsbrekken, PhD, Study Chair — University Hospital, Akershus
Locations (4):
- Norway (4):
  - Akershus University Hospital, Oslo, Lørenskog
  - Vestre Viken HF, Drammen, Vestfold
  - Oslo University Hospital, Oslo
  - Sykehuset Østfold HF, Fredrikstad, Østfold fylke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myhrvold SB, Brouwer EF, Andresen TKM, Rydevik K, Amundsen M, Grun W, Butt F, Valberg M, Ulstein S, Hoelsbrekken SE. Nonoperative or Surgical Treatment of Acute Achilles' Tendon Rupture. N Engl J Med. 2022 Apr 14;386(15):1409-1420. doi: 10.1056/NEJMoa2108447. PMID 35417636

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT01785264/SAP_000.pdf